CLINICAL TRIAL: NCT01673672
Title: A Randomized, Placebo-Controlled, Phase IIb Dose-Finding Study of CYT003-QbG10, a TLR9-Agonist, in Patients With Moderate to Severe Allergic Asthma Not Sufficiently Controlled on Current Standard Therapy (GINA Steps 3+4)
Brief Title: CYT003-QbG10, a TLR9-agonist, for Treatment of Uncontrolled Moderate to Severe Allergic Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: primary endpoint missed
Sponsor: Cytos Biotechnology AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYT003-QbG10 12; 2012-003070-39 (EudraCT Number)
Record Dates: First submitted 2012-08-23; First posted 2012-08-28 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Moderate to Severe Allergic Asthma
MeSH Terms: interventions — CYT003-QbG10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): 7 weekly/biweekly injections of a placebo buffer
  Interventions: Biological: Placebo
- CYT003 low dose (Experimental): 7 weekly/biweekly injections of CYT003 low dose
  Interventions: Biological: CYT003
- CYT003 medium dose (Experimental): 7 weekly/biweekly injections of CYT003 medium dose
  Interventions: Biological: CYT003
- CYT003 high dose (Experimental): 7 weekly/biweekly injections of CYT003 high dose
  Interventions: Biological: CYT003

INTERVENTIONS:
Biological: CYT003 — 7 subcutaneous injections, weekly/biweekly within 10 weeks
  Arms: CYT003 high dose; CYT003 low dose; CYT003 medium dose
Biological: Placebo — 7 subcutaneous injections, weekly/biweekly within 10 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the therapeutic potential and safety/tolerability of study drug (CYT003) at 3 dose levels versus placebo in patients with persistent moderate to severe allergic asthma not sufficiently controlled on current standard controller therapy.

Altogether 360 patients randomized to 4 treatment groups will be included. The study compares three dose strength with placebo. Each patient receives 7 injections of study drug or undistinguishable placebo. Key outcome measures are patient reported parameters on their asthma.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent
* Able and willing to complete all protocol requirements
* Between 18 to 65 years of age
* Presence of persistent asthma for at least 6 months according to GINA 2011 guidelines at step 3 or 4 of treatment who has been on stable controller therapy for at least 4 weeks, and symptoms are not sufficiently controlled with medium to high doses of inhaled corticosteroid (ICS) (>250 to ≤1000 µg/day fluticasone or equivalent) in combination with or without long acting beta agonist (LABA), insufficient control will be based on asthma control questionnaire (ACQ) score ≥1.5 points. Use of stable doses of other controller therapies according to GINA steps 3 and 4 (leukotriene modifiers, sustained release theophylline) are also acceptable, but NOT treatment with anti immunoglobulin E (IgE) antibodies within the past 6 months
* Stable but insufficiently controlled baseline conditions as documented by ACQ ≥1.5 at the screening and the baseline visits.
* Positive skin prick test (SPT) or radioallergosorbent test (RAST) to at least 1 aero-allergen during the screening period
* Forced expiratory volume in one second (FEV1)≥40 to ≤90% of predicted value
* Reversibility of airway obstruction as demonstrated by:

  * FEV1 improvement by >12% , and
  * By ≥200 mL after inhaled β2-agonist (400 µg salbutamol or equivalent). If a subject does not meet reversibility criteria at the screening visit, reversibility may be retested once prior to run-in as long as the test is performed at least 5 days prior to the beginning of the run-in phase

Exclusion Criteria:

* Failure to meet at least 80% compliance with completion of asthma symptoms and medication diaries at the baseline visit, after initial instruction at the screening visit and where necessary additional training at the 2-weeks run-in visit. . An additional maximum 2-weeks training period may be added in such patients.
* Treatment or hospitalization for asthma exacerbation within past 2 months.
* Current use or use of systemic corticosteroids within past 2 months.
* Current smokers.
* Ex-smokers with a smoking history of >10 pack years (1 package per day for 10 years).
* Pregnancy or female planning to become pregnant during the study period.
* Ongoing or planned specific immunotherapy (SIT) during the whole study period or SIT completed within the last 3 years.
* Treatment with IgE antibodies (Xolair®) within past 6 months.
* Use of investigational unapproved drugs within 30 days or within 5 half-lives of the investigational drug, whichever is longer, or planned use during the whole study period.
* Use of investigational biologics within the last 6 months.
* Previous participation in a clinical study with a virus like particle (VLP) Qb-based vaccine.
* Possible dependency of the patient on sponsor and/or investigator.
* Women of child bearing potential

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2012-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Asthma Control Questionnaire | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Casale, Professor, Study Chair — Creighton University, Omaha (NE)
Locations (34):
- United States (21):
  - Cytos Investigator Sites, Los Angeles, Huntington Beach, San Jose, California
  - Cytos Investigator Sites, Walnut Creek, San Diego, Riverside, Fountain Valley, California
  - Cytos Investigator Sites, Colorado Springs, Denver, Colorado
  - Cytos Investigator Sites, Waterbury, Connecticut
  - Cytos Investigator Sites, Miami, Tallahassee, Florida
  - Cytos Investigator Sites, Albany, Georgia
  - Cytos Investigator Sites, South Bend, Indiana
  - Cytos Investigator Sites, Metairie, Louisiana
  - Cytos Investigator Sites, Bangor, Maine
  - Cytos Investigator Sites, Bethesda, Maryland
  - Cytos Investigator Sites, North Dartmouth, Massachusetts
  - Cytos Investigator Sites, St Louis, Missouri
  - Cytos Investigator Sites, Ohmaha, Bellevue, Nebraska
  - Cytos Investigator Sites, Rochester, New York
  - Cytos Investigator Sites, Cincinnati, Ohio
  - Cytos Investigator Sites, Oklahoma City, Oklahoma
  - Cytos Investigator Sites, Eugene, Medford, Oregon
  - Cytos Investigator Sites, Providence, Warwick, Rhode Island
  - Cytos Investigator Sites, Spartanburg, Summerville, South Carolina
  - Cytos Investigator Sites, San Antonio, Texas
  - Cytos Investigator Sites, Richmond, Virginia
- Czechia (2):
  - Cytos Investigator Sites, Kyjov
  - Cytos Investigator Sites, Olomouc, Praha, Tabor, Ostrava, Hradec Kralove, Plzen, Brno
- Germany (2):
  - Cytos Investigator Sites, Bad Woerishofen, Leipzig, Magdeburg
  - Cytos Investigator Sites, Frankfurt aM, Delitzsch, Bonn, Berlin, Ruedersdorf
- Hungary (2):
  - Cytos Investigator Sites, Szazhalombatta, Komaron
  - Cytos Investigator Sites, Tatabanya, Szombathely, Csorna, Budapest, Balassagyarmat
- Israel (2):
  - Cytos Investigator Sites, Haifa, Zerifin
  - Cytos Investigator Sites, Rehovot, Petach Tikva, Ramat Gan, Jerusalem, Ashkelon, Afula
- Cytos Investigator Sites, Slupsk, Lodz, Tarnow, Pila, Poznan, Wroclaw, Poland
- Russia (2):
  - Cytos Investigator Sites, Tomsk,St.Petersburg,Yaroslavl,Novosibirsk,Smolensk,Barnaul
  - Cytos Investigator Sites, Yekaterinburg
- Ukraine (2):
  - Cytos Investigator Sites, Donetsk, Kharkiv, Kiew, Chernivtsi, Zaporizhzhya, Mykolayiv
  - Cytos Investigator Sites, Vinnytsya, Ivano-Frankivsk